CLINICAL TRIAL: NCT05232825
Title: A Study To Investigate The Pharmacokinetics, Pharmacodynamics, Safety And Radiological And Clinical Effects Of Subcutaneous Ocrelizumab Versus Intravenous Ocrelizumab In Patients With Multiple Sclerosis
Brief Title: A Phase III, Non-Inferiority, Randomized, Open-Label, Parallel Group, Multicenter Study To Investigate The Pharmacokinetics, Pharmacodynamics, Safety And Radiological And Clinical Effects Of Subcutaneous Ocrelizumab Versus Intravenous Ocrelizumab In Patients With Multiple Sclerosis
Acronym: Ocarina II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CN42097
Record Dates: First submitted 2022-01-27; First posted 2022-02-10 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Relapsing Multiple Sclerosis; Primary Progressive Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ocrelizumab: Intravenous (IV) formulation (Active Comparator): Participants will receive the first dose of ocrelizumab IV as two IV infusions given 14 days apart. The subsequent doses of study drug will be administered as SC injections. A minimum of 22 weeks should be kept between SC doses. Participants will undergo 96 weeks of study treatment.
  Interventions: Drug: Ocrelizumab IV; Drug: Methylprednisolone IV; Drug: Diphenhydramine IV
- Ocrelizumab: Subcutaneous (SC) formulation (Experimental): Participants will receive the first dose of ocrelizumab SC as one SC injection at a dose which is expected to result in non-inferior exposure to ocrelizumab IV. The subsequent doses of study drug will be administered as SC injections. A minimum of 22 weeks should be kept between the first and second SC doses, and between subsequent SC doses. Participants will undergo 96 weeks of study treatment.
  Interventions: Drug: Ocrelizumab SC; Drug: Dexamethasone given orally; Drug: Desloratadine given orally

INTERVENTIONS:
Drug: Ocrelizumab IV — IV Injection
  Other Names: RO4964913
  Arms: Ocrelizumab: Intravenous (IV) formulation
Drug: Ocrelizumab SC — SC Injection
  Other Names: RO4964913
  Arms: Ocrelizumab: Subcutaneous (SC) formulation
Drug: Methylprednisolone IV — Participants will receive mandatory (corticosteroids and antihistamine) and optional (analgesic) prophylactic treatment before the start of each ocrelizumab infusion
  Arms: Ocrelizumab: Intravenous (IV) formulation
Drug: Diphenhydramine IV — Participants will receive mandatory (corticosteroids and antihistamine) and optional (analgesic) prophylactic treatment before the start of each ocrelizumab infusion
  Arms: Ocrelizumab: Intravenous (IV) formulation
Drug: Dexamethasone given orally — Participants will receive mandatory (corticosteroids and antihistamine) and optional (analgesic) prophylactic treatment before the start of each ocrelizumab injection
  Arms: Ocrelizumab: Subcutaneous (SC) formulation
Drug: Desloratadine given orally — Participants will receive mandatory (corticosteroids and antihistamine) and optional (analgesic) prophylactic treatment before the start of each ocrelizumab injection
  Arms: Ocrelizumab: Subcutaneous (SC) formulation

SUMMARY:
This study will evaluate the pharmacokinetics, pharmacodynamics, safety, immunogenicity, and radiological and clinical effects of subcutaneous (SC) administration of ocrelizumab compared with the intravenous (IV) infusion of ocrelizumab in patients with either relapsing multiple sclerosis (RMS) or primary progressive multiple sclerosis (PPMS).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PPMS or RMS according to the revised McDonald 2017 criteria (Thompson et al. 2018)
* EDSS score, 0-6.5, inclusive, at screening
* Neurological stability for ≥30 days prior to both screening and baseline
* Disease duration from onset of MS symptoms of less than 15 years for patients with EDSS score <2.0 at screening
* For females participants, without reproductive potential may be enrolled if post-menopausal, unless receiving a hormonal therapy for menopause or if surgically sterile
* For females of childbearing potential, agreement to remain abstinent or use adequate contraceptive methods

Exclusion Criteria:

* Any known or suspected active infection at screening or baseline (except nailbed infections), or any major episode of infection requiring hospitalization or treatment with IV anti microbials within 8 weeks prior to and during screening or treatment with oral anti microbials within 2 weeks prior to and during screening
* History of confirmed or suspected progressive multifocal leukoencephalopathy (PML)
* History of cancer, including hematologic malignancy and solid tumors, within 10 years of screening
* Immunocompromised state
* Receipt of a live-attenuated vaccine within 6 weeks prior to randomization Influenza vaccination is permitted if the inactivated vaccine formulation is administered
* Inability to complete an MRI or contraindication to gadolinium administration
* Contraindications to mandatory premedications for IRRs, including closed-angle glaucoma for antihistamines
* Known presence of other neurologic disorders
* Any concomitant disease that may require chronic treatment with systemic corticosteroids or immunosuppressants during the course of the study
* Significant, uncontrolled disease, such as cardiovascular, pulmonary, renal, hepatic, endocrine or gastrointestinal, or any other significant disease that may preclude patient from participating in the study
* History of or currently active primary or secondary (non-drug-related) immunodeficiency
* Pregnant or breastfeeding, or intending to become pregnant during the study and 6 or 12 months
* Lack of peripheral venous access
* History of alcohol or other drug abuse within 12 months prior to screening
* Treatment with any investigational agent within 24 weeks prior to screening or 5 half-lives of the investigational drug (whichever is longer), or treatment with any experimental procedure for MS (e.g., treatment for chronic cerebrospinal venous insufficiency)
* Participants who have previously received anti-CD20s if the last treatment was less than 2 years before screening, and/or if B-cell count is below lower limit of normal, and/or the discontinuation of the treatment was due to safety reasons or lack of efficacy
* Previous treatment with cladribine, atacicept, and alemtuzumab
* Previous treatment with fingolimod, siponimod, ponesimod, or ozanimod within 6 weeks of baseline
* Previous treatment with interferons beta (1a or 1b), or glatiramer acetate within 2 weeks of baseline
* Previous treatment with natalizumab within 4.5 months of baseline
* Treatment with mitoxantrone within 2 years prior to baseline visit or evidence of cardiotoxicity following mitoxantrone use or a cumulative lifetime dose of more than 60 mg/m2
* Previous treatment with any other immunomodulatory or immunosuppressive medication not already listed above without appropriate washout as described in the applicable local label.
* If the washout requirements are not described in the applicable local label, then the wash out period must be 5 times the half-life of the medication. The PD effects of the previous medication must also be considered when determining the required time for washout.
* Any previous treatment with bone marrow transplantation and hematopoietic stem cell transplantation
* Any previous history of transplantation or anti-rejection therapy
* Treatment with IV Ig or plasmapheresis within 12 weeks prior to randomization
* Systemic corticosteroid therapy within 4 weeks prior to screening
* Positive screening tests for active, latent, or inadequately treated hepatitis B
* Sensitivity or intolerance to any ingredient (including excipients) of ocrelizumab
* Any additional exclusionary criterion as per ocrelizumab (Ocrevus®) local label, if more stringent than the above

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2022-05-03 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2025-06-06 (Actual)

PRIMARY OUTCOMES:
Serum ocrelizumab area under the concentration-time curve (AUCW1-12) | Day 1 to Week 12

SECONDARY OUTCOMES:
Maximum serum concentration (Cmax) of ocrelizumab SC in patients with MS | Day 1 to Week 12
Total number of T1Gd+ lesions as detected by brain MRI | Weeks 8 and 24
Total number of new or enlarging T2 lesions as detected by brain MRI | Weeks 12 and 24
Percentage of participants with Adverse Events | Day 1 to Week 48
Incidence of treatment-emergent antidrug antibodies to ocrelizumab after SC or IV administration | Day 1 to Week 48
Incidence of treatment-emergent antibodies to rHuPH20 | Day 1 to Week 48
Proportion of participants achieving CD19+ B cell level ≤5 cells/uL | Day 1 to Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (37):
- United States (7):
  - Neurology Associates PA, Maitland, Florida
  - University of South Florida, Tampa, Florida
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Memorial Healthcare Institute for Neurosciences and Multiple Sclerosis, Owosso, Michigan
  - UC Health Neurology, Dayton, Ohio
  - Premier Neurology, Greenville, South Carolina
  - Neurology Clinic PC, Cordova, Tennessee
- Brazil (2):
  - CEDOES - Diagnóstico e Pesquisa, Vitória, Espírito Santo
  - Clinica Amo - Assistencia Medica Em Oncologia, Salvador, Estado de Bahia
- Czechia (8):
  - Fakultni nemocnice u sv. Anny, Brno
  - Charles University, Medical faculty, Hradec Kralove, Hradec Králové
  - Nemocnice Jihlava, Jihlava
  - Fakultni nemocnice Ostrava, Ostrava-Poruba
  - Pardubicka Krajska Nemocnice, Pardubice
  - Fakultni poliklinika VFN, Prague
  - Fakultni nemocnice Motol, Prague
  - Krajska zdravotni a.s Nemocnice Teplice o.z., Teplice
- Italy (4):
  - Policlinico Tor Vergata Dip. Neuroscienze-Clinica Neurologica-UOSD Sclerosi Multipla, Rome, Lazio
  - Azienda Ospedaliera Sant'Andrea, Rome, Lazio
  - Ospedale Civile di Montichiari, Montichiari, Lombardy
  - IRCCS Istituto Neurologico Neuromed, Pozzilli, Molise
- New Zealand (2):
  - Optimal Clinical Trials, Auckland
  - Hawkes Bay Hospital, Hastings
- Poland (4):
  - Neurocentrum Bydgoszcz sp. z o.o, Bydgoszcz
  - Care Clinic, Katowice
  - Centrum Neurologii Krzysztof Selmaj, Lodz
  - Przychodnia EuroMediCare, Wroc?aw
- Spain (5):
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital Universitario Virgen Macarena, Seville, Sevilla
  - Complejo Hospitalario Nuestra Señora de la Candelaria, Santa Cruz de Tenerife, Tenerife
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
- Turkey (Türkiye) (5):
  - Bakirkoy State Mental Hospital, Istanbul
  - Istanbul Universitesi - Cerrahpasa Cerrahpasa Tip Fakultesi, Istanbul
  - Katip Celebi University Ataturk Training and Research Hospital, Izmir
  - Kocaeli University Hospital, Kocaeli
  - Namik Kemal Universitesi Sagli Uygulama ve Arastirma Hastanesi, Süleymanpa?a

REFERENCES:
- [Derived] Newsome SD, Krzystanek E, Selmaj KW, Dufek M, Goldstick L, Pozzilli C, Figueiredo C, Townsend B, Kletzl H, Bortolami O, Zecevic D, Giacobino C, Clinch S, Shen YA, Bhullar GD, Schneble HM, Centonze D. Subcutaneous Ocrelizumab in Patients With Multiple Sclerosis: Results of the Phase 3 OCARINA II Study. Neurology. 2025 May 13;104(9):e213574. doi: 10.1212/WNL.0000000000213574. Epub 2025 Apr 17. PMID 40245351
- [Derived] Newsome SD, Goldstick L, Robertson DS, Bowen JD, Naismith RT, Townsend B, Figueiredo C, Kletzl H, Giraudon M, Bortolami O, Zecevic D, Giacobino C, Clinch S, Shen YA, Deol-Bhullar G, Bermel RA. Subcutaneous ocrelizumab in multiple sclerosis: Results of the Phase 1b OCARINA I study. Ann Clin Transl Neurol. 2024 Dec;11(12):3215-3226. doi: 10.1002/acn3.52229. Epub 2024 Oct 26. PMID 39460719